CLINICAL TRIAL: NCT02711735
Title: Double-Blind, Randomized, Placebo-Controlled Phase IIa Clinical Trial to Investigate the Safety and Immunogenicity of RUTI® Therapeutic Vaccination in Patients With MDR-TB After Successful Intensive-phase Treatment.
Brief Title: Safety of RUTI® Vaccination in MDR-TB Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Archivel Farma S.L. (Industry)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201600136; 2016-000850-36 (EudraCT Number)
Record Dates: First submitted 2016-02-25; First posted 2016-03-17 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Tuberculosis, Multidrug Resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUTI® vaccine (Active Comparator): Intervention: Patients randomized to receive RUTI® vaccine will receive one injection of RUTI® vaccine in their right or left deltoid muscle.
  Interventions: Biological: RUTI® Therapeutic vaccine
- Matching RUTI® Placebo (Placebo Comparator): Intervention: Patients randomized to receive Placebo will receive one injection of Placebo in their right or left deltoid muscle.
  Interventions: Biological: Matching RUTI® Placebo

INTERVENTIONS:
Biological: RUTI® Therapeutic vaccine — Participants randomised to this arm will receive one single dose of RUTI® vaccine in the right/left deltoid muscle.
  Arms: RUTI® vaccine
Biological: Matching RUTI® Placebo — Participants randomised to this arm will receive aone single dose of matching RUTI® placebo in the right / left deltoid
  Arms: Matching RUTI® Placebo

SUMMARY:
Prospective, randomized, double-blind, multicentre, placebo-controlled clinical phase IIa trial to evaluate safety and immunogenicity of RUTI® vaccine in Multidrug-resistant Tuberculosis (MDR-TB) patients favourably responding to standard MDR-TB treatment. Time point of vaccination starts at 16 weeks upon start of standard MDR-TB treatment (cohort A), and if clinically safe as evaluated by an independent panel of experts (DSMB), another cohort of patients will be vaccinated at 2 weeks upon start of standard MDR-TB treatment (cohort B), All the patients will be followed up 8 weeks after vaccination.

DETAILED DESCRIPTION:
Prospective, randomized, double-blind, multicentre, placebo-controlled clinical phase IIa trial to evaluate safety and immunogenicity of RUTI® vaccine in Multidrug-resistant Tuberculosis (MDR-TB) patients favourably responding to standard MDR-TB treatment. Time point of vaccination starts at 16 weeks upon start of standard MDR-TB treatment (cohort A), and if clinically safe as evaluated by an independent panel of experts (DSMB), another cohort of patients will be vaccinated at 2 weeks upon start of standard MDR-TB treatment (cohort B)

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Diagnosed with pulmonary MDR-TB, and therefore managed with second line TB drugs;
* Admitted in a TB unit / hospital routinely diagnosed with pulmonary MDR-TB with clinical status ≥ 6 with Bandim TB score combined with chest radiography; and microbiological criteria according to the medical history), using rapid genetic testing (GeneXpert TB test) and MGIT to confirm or Line Probe Assay; or classical diagnostic tools including sputum microscopy and culture followed by phenotypic drug susceptibility testing. All of this medical information will be in the medical history;
* Females and males aged ≥ 18; females of non-childbearing potential: at least 2 years post-menopausal or surgically sterile (e.g. tubal ligation); females of childbearing potential (including females less than 2 years post-menopausal) must have a negative pregnancy test at enrolment and must agree to use highly effective methods of birth control (i.e. diaphragm plus spermicide or male condom plus spermicide, oral contraceptive in combination with a second method, contraceptive implant, injectable contraceptive, indwelling intrauterine device, sexual abstinence, or a vasectomized partner) while participating in the study and for 30 days after end of the study for each group; males must agree to use a double barrier method of contraception (condom plus spermicide or diaphragm plus spermicide) while participating in the study and for 30 days after end of the study for the respective group; or the male patient or his female partner must be surgically sterile (e.g. vasectomy, tubal ligation) or the female partner must be post-menopausal;
* The patient must provide written informed consent;
* The patient must be willing and able to attend all study visits and comply with all study procedures.

Inclusion criteria for vaccination

* Having successfully completed 16, 8 or 4 weeks (depending on the cohort) of MDR-TB treatment, fully supervised, and
* With beneficial initial response to therapy, evidenced by:

Clinical response criteria: patients admitted in a TB unit / hospital routinely diagnosed with pulmonary MDR-TB (according to clinical status ≤ 5 with Bandim TB score) (33).

Transient deterioration of chest radiographic abnormalities might be explained by a paradoxical inflammatory response, and this may therefore not necessarily be interpreted as treatment failure; such decision depends on consensus with the DSMB; evidence of improvement on chest x-ray.

• Microbiological response criteria: It has to be reported a reduction of the bacillary load in the sputum by means of the reduction of bacillary counts in GeneXpert TB test and liquid culture (MGIT) to confirm (diagnosis week 0 collected in the medical history) at week 4 in CohortsC, week 8 in both Cohorts (A-B) and week 12 and 16 in Cohort A.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Inability to provide written informed consent;
* Women reported, or detected, or willing to be pregnant during the trial period;
* Severity of illness precluding full evaluation: expected early death, evidenced by respiratory failure, low blood pressure, WHO performance score 3-4; Central Nervous System involvement of TB (TB meningitis, intra-cranial tuberculomas) as there is too little evidence for effective drug penetration for second-line TB drugs;
* Major co-morbid conditions precluding full evaluation, i.e., active lung cancer, acute coronary syndrome, heart failure exceeding NYHA class 2; a diagnosis of metastasized malignancy; renal failure in excess of creatinine clearance < 30 mL/min calculated by the Cockcroft-Gault formula, which would severely complicate administration of aminoglycosides and capreomycin, considered as the major second-line TB drugs; obesity (BMI>30 kg/m2); chronic liver disease - Child-Pugh class C;
* Any of the following laboratory parameters:

Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN) Total bilirubine > 2 x ULN Neutrophil count ≤ 500 neutrophils / mm3 Platelet count < 50,000 cells / mm3

* Receiving or anticipated to receive a daily dose of ≥ 10 mg of systemic prednisone or equivalent within the period starting 14 days prior to enrolment. Note: patients are allowed to receive an acute, short course of methylprednisolone or prednisone or equivalent for management of an acute exacerbation of COPD or reactive airway disease in asthmatics;
* Cytotoxic chemotherapy or radiation therapy within the previous 3 months;
* HIV co-infection, if CD4 count < 250 cells/mm3 at the diagnosis of HIV; those with > 250 copies/mL are expected to be able to mount a sufficient cellular immune response and will therefore be eligible;
* Blood transfusion in the last three weeks prior to the trial;
* Documented allergy to TB vaccines, notably, to the RUTI® vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Clinical safety parameters related to vaccination | 8 weeks
  Safety Evaluation: Physical examination, SAEs, routine laboratory, chest radiography, between the intervention and control group within 8 weeks after vaccination.

SECONDARY OUTCOMES:
IFN-y release of PBMCs in response to antigen stimulation | 8 weeks
  Immunogenicity Evaluation: Immunogenic properties of RUTI® vaccine (before vaccination and at week 2 and 8 after vaccination) compared to placebo assessed by i) IFN-γ production of ex vivo stimulated peripheral blood mononuclear cells (PBMC)
Mycobacterial Growth Inhibition Assay | 8 weeks
  Immunogenicity Evaluation: Immunogenic properties of RUTI® vaccine (before vaccination and at week 2 and 8 after vaccination) compared to placebo assessed by the summative ability of PBMCs to control mycobacterial growth in an ex vivo system.

CONTACTS AND LOCATIONS:
Overall Officials: Tjip S van der Werf, MD PhD, Principal Investigator — University Medical Center Groningen, The Netherlands
Locations (3):
- Ukraine (3):
  - "Chernivtsi Regional Clinical TB Dispensary", II tuberculosis department of multidrug-resistant tuberculosis, Chernivtsi
  - "Ivano-Frankivsk Regional Phthisiopulmonology Center of Ivano-Frankivsk Regional Council", Center for Pulmonary Diseases, Ivano-Frankivsk
  - Medical Department #2 (resistant tuberculosis) of Kharkiv Regional Antituberculosis Dispensary No1, Kharkiv

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Vilaplana C, Montane E, Pinto S, Barriocanal AM, Domenech G, Torres F, Cardona PJ, Costa J. Double-blind, randomized, placebo-controlled Phase I Clinical Trial of the therapeutical antituberculous vaccine RUTI. Vaccine. 2010 Jan 22;28(4):1106-16. doi: 10.1016/j.vaccine.2009.09.134. Epub 2009 Oct 22. PMID 19853680
- [Background] Nell AS, D'lom E, Bouic P, Sabate M, Bosser R, Picas J, Amat M, Churchyard G, Cardona PJ. Safety, tolerability, and immunogenicity of the novel antituberculous vaccine RUTI: randomized, placebo-controlled phase II clinical trial in patients with latent tuberculosis infection. PLoS One. 2014 Feb 26;9(2):e89612. doi: 10.1371/journal.pone.0089612. eCollection 2014. PMID 24586912